CLINICAL TRIAL: NCT03380026
Title: Valchlor Therapy in Conjunction With Triamcinolone 0.1% Ointment for the Treatment of Contact Dermatitis in Patients With Early Stage Cutaneous T-cell Lymphoma (Mechlorethamine Induced Dermatitis Avoidance Study)
Brief Title: Mechlorethamine Induced Contact Dermatitis Avoidance Study
Acronym: MIDAS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rochester Skin Lymphoma Medical Group, PLLC (Other)
Collaborators: Rochester General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RSLMG-17.10
Record Dates: First submitted 2017-12-12; First posted 2017-12-20 (Actual); Results first posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-10

CONDITIONS: Cutaneous T-cell Lymphoma; Cutaneous T-cell Lymphoma Stage I; Mycosis Fungoides; Folliculotropic Mycosis Fungoides; Granulomatous Slack Skin; Syringotropic Mycosis Fungoides; Mycosis Fungoides Variant; Transformed Mycosis Fungoides
Keywords: CTCL; topical mechlorethamine; Valchlor; contact dermatitis; triamcinolone; MF; Cutaneous T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Dermatitis, Contact | interventions — Triamcinolone; Triamcinolone Acetonide; Ointments; Amines; Gels; Mechlorethamine

STUDY DESIGN:
Intervention Model Description: open-label, split-face study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Valchlor 0.016% Topical Gel (Experimental): 0.016% w/w topical mechlorethamine gel applied over a minimum of 8 cm2, nightly, over a period of 4 months.
  Interventions: Drug: Valchlor 0.016 % Topical Gel
- Valchlor plus Triamcinolone (Active Comparator): 0.016% w/w topical mechlorethamine gel (once, nightly) and Triamcinolone acetonide 0.1% ointment (up to three times daily) applied in over a minimum of 8 cm2, over a period of 4 months.
  Interventions: Drug: Triamcinolone; Drug: Valchlor 0.016 % Topical Gel

INTERVENTIONS:
Drug: Triamcinolone — Apply up to three times daily on select lesions.
  Other Names: triamcinolone acetonide; Triamcinolone 0.1% ointment
  Arms: Valchlor plus Triamcinolone
Drug: Valchlor 0.016 % Topical Gel — Apply valchlor nightly on select lesions.
  Other Names: topical nitrogen mustard; mechlorethamine hydrochloride; mechlorethamine gel

SUMMARY:
This is a two-arm, open-label study that aims to compare the incidence and severity of the most common adverse reactions, particularly contact dermatitis, when Valchlor is used alone or in conjunction with triamcinolone ointment 0.1% in early stage MF subjects (Stage IA and IB) for a period of 4 months.

DETAILED DESCRIPTION:
Mechlorethamine hydrochloride, or most commonly known as nitrogen nitrogen mustard, was approved by the FDA in 2013 for the treatment of IA and IB Mycosis Fungoides. The most common side effect of Valchlor is a skin rash, which is routinely ameliorated with the application of topical corticosteroids, such as topical Triamcinolone. The main purpose of this study is to determine the efficacy of Triamcinolone in reducing side effects cause by Valchlor and further understand the nature of this skin rash.

This is a split-face study, meaning that subjects will receive both therapies, but limit use to designated areas. Treatment lasts 4 months with follow ups at 5 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Be eligible to receive Valchlor therapy.
* Be at least of 18 years of age and ability to give informed consent
* Have stage IA or IB CTCL
* Subjects with histologic variants of Mycosis Fungoides such as folliculotropic, granulomatous slack skin, syringotropic MF, or large cell transformation ARE eligible.
* A skin biopsy within the last 60 days before start of treatment. In cases with equivocal histological features, the diagnosis may be confirmed with clinicopathologic and/or genetic testing consistent with the National Comprehensive Cancer Network guidelines for Mycosis Fungoides. If sufficient tissue is not available to perform genetic testing, a new biopsy will be performed even if the subject has had a biopsy within 60 days of start of treatment.
* Females of child bearing potential must agree to use two highly effective methods of contraception (strongly recommended that one of the two forms of contraception be non-hormonal such as condom plus spermicide, condom plus diaphragm with spermicide, or have a vasectomized partner) or use an intrauterine device until 30 days after the last day of drug administration. Perimenopausal women must be amenorrhoeic for at least 12 months to be considered of nonchildbearing potential.
* Males with female partners of child bearing potential must agree to sexual abstinence or use two reliable forms of effective contraception simultaneously (strongly recommended that one of the two forms should be non-hormonal as described above) during the entire treatment period and 30 days after the last dose.
* Must be able to comply with the study instructions, apply the study medication as directed, and attend all visits.
* Willingness to avoid sun exposure and ultraviolet B light in areas to be treated.

Exclusion Criteria:

* Have been treated with topical mechlorethamine within 6 months in lesions followed during this study.
* Have received any topical therapy directed against MF within 2 weeks of start of treatment in areas intended to be treated in this study.
* Have received any systemic therapy (oral or injectables) within 3 weeks of start of treatment.
* Not have any intercurrent illness or infection that would interfere with study participation
* Known hypersensitivity to mechlorethamine or triamcinolone.
* Breastfeeding, pregnancy, or intention to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2020-08-03 (Actual); Study Completion 2020-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Poligone, MD, PhD, Principal Investigator — Rochester Skin Lymphoma Medical Group, PLLC
Locations (1):
- Rochester Skin Lymphoma Medical Group, PLLC, Fairport, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be embargoed until the study site has fully examined it. Expected embargo would be one year from study completion.
  Study data that is de-identified will be maintained at the study site. As this field is rapidly changing, if a database is available for safe, public upload at the end of study embargo, it will be uploaded to a national database. Otherwise requests for use of the study data will be accepted at the study site and shared with investigators whose proposed use of data has been approved by an independent institutional review board. Contact addresses and phone numbers will be presented on all publications to assist in this study sharing.
Supporting Information: CSR
Time Frame: Expected embargo would be one year from study completion. De-identified data will be maintained at the study site for 2 years after the study ends. Contact addresses and phone numbers will be presented on all publications to assist in this study sharing.
Access Criteria: Data will be shared with investigators whose proposed use of data has been approved by an independent institutional review board.

REFERENCES:
- [Background] Lessin SR, Duvic M, Guitart J, Pandya AG, Strober BE, Olsen EA, Hull CM, Knobler EH, Rook AH, Kim EJ, Naylor MF, Adelson DM, Kimball AB, Wood GS, Sundram U, Wu H, Kim YH. Topical chemotherapy in cutaneous T-cell lymphoma: positive results of a randomized, controlled, multicenter trial testing the efficacy and safety of a novel mechlorethamine, 0.02%, gel in mycosis fungoides. JAMA Dermatol. 2013 Jan;149(1):25-32. doi: 10.1001/2013.jamadermatol.541. PMID 23069814
- [Derived] Alexander-Savino CV, Chung CG, Gilmore ES, Carroll SM, Poligone B. Randomized Mechlorethamine/Chlormethine Induced Dermatitis Assessment Study (MIDAS) Establishes Benefit of Topical Triamcinolone 0.1% Ointment Cotreatment in Mycosis Fungoides. Dermatol Ther (Heidelb). 2022 Mar;12(3):643-654. doi: 10.1007/s13555-022-00681-6. Epub 2022 Feb 5. PMID 35122614
- See also: Valchlor package insert — https://www.accessdata.fda.gov/drugsatfda_docs/label/2013/202317lbl.pdf
- See also: Triamcinolone acetonide information — https://dailymed.nlm.nih.gov/dailymed/archives/fdaDrugInfo.cfm?archiveid=12961

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients presenting to medical clinic eligible for mechlorethamine topical therapy.
Pre-assignment Details: Two week wash out. Prior to treatment, one half of each patient's body (divided sagittally at the midline) is assigned to treatment with Valchlor only, while the other side of the patient's body is assigned to treatment with both Valchlor and Triamcinolone Acetonide. Group assignment is determined randomly by the flip of a coin.
Groups:
- All Participants: Group consisting of all trial participants that completed screening and randomization.
  In this split-person study, lesions from one half of each participant's body are assigned to one of two treatment groups: One half of the body is assigned to treatment of affected lesions with Valchlor only, while the other half of the body is assigned to treatment of affected lesions with both Valchlor and Triamcinolone.
  For the Valchlor only group, Valchlor is applied once nightly to the target lesions.
  For the Valchlor + Triamcinolone group, 0.016% w/w topical mechlorethamine gel is applied once nightly to target lesions, and Triamcinolone acetonide 0.1% ointment is applied up to three time per day to target lesions over a minimum of 8 cm2
  For both groups, the treatment period spanned four months.
Period: Overall Study
Arm/Group | All Participants
Started | 28
Half of Body Assigned to Treatment With Valchlor Only (Side of body from each patient assigned to treatment with Valchlor only, assigned randomly at enrollment.) | 28
Half of Body Assigned to Treatment With Valchlor and Triamcinolone Acetonide (Side of body from each patient assigned to treatment with both Valchlor and Triamcinolone, assigned randomly at enrollment.) | 28
Completed | 25
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 28
Age, Customized [Count of Participants; unit: Participants]
  21-30 | 2
  31-40 | 1
  41-50 | 2
  51-60 | 6
  61-70 | 7
  71-80 | 7
  81-90 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Moderate to Severe Contact Dermatitis by SCORD Scoring
Description: Incidence of moderate to severe contact dermatitis in patients treated concurrently with Triamcinolone 0.1% ointment versus those that are not. Dermatitis will be defined as a finding of cutaneous inflammatory reaction occurring as a result of treatment. This will be assessed by the SCORD (SCORing Dermatitis) tool and may be confirmed by biopsy of the specimen. Moderate to Severe Contact dermatitis is defined as >25 by SCORD.
Time Frame: 4 months
Population: Each patient had both treatments (self-controlled)
Measure: Number; unit: patients
Arm/Group | Valchlor 0.016% Topical Gel | Valchlor Plus Triamcinolone
Number analyzed (Participants) | 27 | 27
patients | 16 | 11

2. Secondary Outcome: Nature of Contact Dermatitis (Allergic Versus Irritant)
Description: The presence of allergic versus irritant dermatitis was characterized through skin biopsies sent for pathological review and patch testing. Subjects presenting to the clinic with dermatitis underwent patch testing to determine the presence of allergic vs. Irritant contact dermatitis, and at each case a biopsy sample was taken of the affected area to confirm the diagnosis. Patch testing was assessed by the investigator according to the International Contact Dermatitis Research Group scale, using the following for possible outcomes : ?+ indicates a doubtful reaction, 1+ indicates a weak reaction, 2+ represents a strong reaction, 3+ indicates an extreme reaction, and IR indicates an Irritant reaction. A higher score would indicate a worse outcome. 1-3+ reaction at the 96hr reading was considered positive for allergic contact dermatitis.
Time Frame: 4 months
Population: All analyzed trial participants Were included in assessment of dermatitis. 12 incidents of dermatitis were observed across the study, and at each incident a biopsy of the affected area was sent for histopathological review. 10 of 12 patients presented with allergic contact dermatitis, while 2 out of 10 12 patients presented with irritant contact dermatitis according to pathology results.
Measure: Count of Units; unit: Incidents of dermatitis
Units Other Than Participants: Incidents of dermatitis
Groups:
- All Participants: Group of all analyzed study participants. Both irritant and allergic contact dermatitis was observed
Arm/Group | All Participants
Number analyzed (Participants) | 27
Number analyzed (Incidents of dermatitis) | 12
Incidents of dermatitis
  Incidents of Contact Dermatitis | 2
  Incidents of Allergic Dermatitis | 10

3. Other Pre Specified Outcome: Severity of Dermatitis
Description: Scoring Atopic Dermatitis (SCORAD) differences between lesions treated with Valchlor and Triamcinolone versus lesions treated with Valchlor only. SCORAD measures the extent and severity of dermatitis. The percentage of total body surface area (0-100) covered by a lesion is measured by an investigator, and this number corresponds to score "A." The intensity criteria are met by scoring erythema, edema/papulation, oozing/crusting, excoriation, xerosis, and thickness on a scale of 0-3 (0=none, 1=mild, 2=Moderate, 3=Severe). These values are summed to give a total score, "B." Subjective symptoms of pruritus and insomnia are then scored using visual analogue scales ranging from 0-10 (0=none, 10=worst imaginable), and the result of each is summed to give score "C". The final score is then calculated by the formula A/5 + 7B/2 + C. The lowest possible score is 0, and the highest possible score is 103. A higher score indicates a worse outcome.
  A lower score would be a better outcome.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Valchlor 0.016% Topical Gel | Valchlor Plus Triamcinolone
Number analyzed (Participants) | 27 | 27
score on a scale | 24.8 (21.8) | 12.7 (13.5)

4. Other Pre Specified Outcome: Efficacy of Valchlor vs Valchlor Plus Triamcinolone
Description: Efficacy of Valchlor therapy with Triamcinolone compared to Valchlor using a composite assessment of index lesion severity (CAILS). CAILS is an objective, quantitative, method to assess the extent of skin lesions. Skin lesions and erythema will be evaluated using CAILS. A Composite Assessment will be generated for each time point by a summation of the grades for each index lesion's erythema, scaling, plaque elevation, hypopigmentation or hyperpigmentation, and area of involvement. The index lesion grade at baseline will be divided into the grade at each subsequent study visit to determine the subject's response to treatment. Any ratio of the grade obtained at the visit vs. the one obtained at baseline that is >1.0 will indicate worsening of disease.
Time Frame: 4 months
Population: CAILS
Measure: Mean (Standard Deviation); unit: CAILS score
Arm/Group | Valchlor 0.016% Topical Gel | Valchlor Plus Triamcinolone
Number analyzed (Participants) | 27 | 27
CAILS score
  Average CAILS score at Baseline | 8.6 (4.2) | 7.0 (5.1)
  Average CAILS score at Month 4 | 11.4 (4.9) | 12.0 (4.85)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Valchlor 0.016% Topical Gel | Valchlor Plus Triamcinolone
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 16/28 | 11/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Valchlor 0.016% Topical Gel (N=28) | Valchlor Plus Triamcinolone (N=28)
Contact Dermatitis (Skin and subcutaneous tissue disorders) | 16 (16) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-11): https://cdn.clinicaltrials.gov/large-docs/26/NCT03380026/Prot_SAP_000.pdf